CLINICAL TRIAL: NCT06242028
Title: Use of Dexamethasone Via Two Different Methods in PENG Block for Patients Undergoing Femoral Fracture Surgery
Brief Title: Use of Dexamethasone Via Two Different Methods in PENG Block
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ebru Kelsaka, Professor Doctor, Ondokuz Mayıs University
Other Study IDs: PENDEX2022
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pain, Acute; Postoperative Pain; Hip Fractures
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P (Perinuerally): Ultrasound guided PENG block with perinuerally dexamethasone administration group
  Interventions: Drug: Group P
- Group S (Systematic): Ultrasound guided PENG block with systemic dexamethasone administration group
  Interventions: Drug: Group S

INTERVENTIONS:
Drug: Group P — In this group, US guided PENG block will be performed with 20 cc 0.25% bupivacaine and 4 mg dexamethasone.
  Other Names: Perinuerally
  Groups: Group P (Perinuerally)
Drug: Group S — In this group, US guided PENG block will be performed with 20 cc 0.25% bupivacaine. In addition, 4 mg dexamethasone will be administered intravenously.
  Other Names: Systematic
  Groups: Group S (Systematic)

SUMMARY:
Hip fractures are morbid conditions, especially in elderly patients, and their treatment is usually surgical. Pericapsular nerve group block targets the hip capsule. The aim of this study is to investigate and compare the perioperative analgesic efficacy of PENG blocks applied investigation of the effect of perinuerally and systemic dexamethasone on pain scores in the first 24 hours of PENG block in patients undergoing hip fracture surgery under spinal anesthesia.

DETAILED DESCRIPTION:
Hip fractures are morbid conditions, especially in elderly patients, and their treatment is usually surgical. Pericapsular nerve group block targets the hip capsule. The aim of this study is to investigate and compare the perioperative analgesic efficacy of PENG blocks applied investigation of the effect of perinuerally and systemic dexamethasone on pain scores in the first 24 hours of PENG block in patients undergoing hip fracture surgery under spinal anesthesia.

44 ASA II-IV patients between 50-80 years of age who will be operated for femoral neck fractures will be included in the study.

PENG block is routinely used in our clinic to provide postoperative analgesia in hip surgery. Depending on the comorbid conditions of the patients, dexamethasone may be added as an adjuvant agent to improve the quality of the block. We aimed to observe the systemic and perinuerally effects of dexamethasone used in PENG block in patients operated for femoral neck fracture in our clinic.

In this observational and prospective study, patients operated for femoral neck fracture and treated with PENG block will be analyzed in the postoperative period. Pain scores, degree of nausea and vomiting, recovery time of sensory and motor block, and blood glucose levels in the first 24 hours will be recorded in patients who received dexamethasone perinuerally and in patients who received systemic dexamethasone intravenously. In addition, the time to first analgesic requirement, mobilization time and hospital stay of the two groups will also be recorded.

The anesthesiologist performing the block will not participate in the pain monitoring of the patients. Postoperative pain assessment and data collection will be performed by another anesthesiologist blinded to the study. For the quality and standardization of the block, the block will be performed by an experienced anesthesiologist who has performed the block successfully and without complications at least 20 times before.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 years old
* Patients who underwent surgery for femoral neck fracture under spinal anesthesia with PENG block
* Patients of either sex with a body mass index (BMI) < 35 kg/m2
* ASA II-IV patients
* Patients signing the informed consent form

Exclusion Criteria:

* ASA-V patients
* Alcohol, drug addiction
* Patients with a history of opioid drug use for more than four weeks
* Patients with chronic pain disorders (patients on regular analgesics >3 months)
* Patients with a history of local anesthetic or opioid allergy or hypersensitivity
* Patient group in whom regional anesthesia is contraindicated (coagulopathy, INR (international correction ratio) not within normal limits, thrombocytopenia or platelet dysfunction, infection at the injection site)
* Those with severe psychiatric illnesses such as psychosis, dementia, etc. that limit their cooperation with the patient
* Patients who do not give consent/ do not want to participate
* Patients who were evaluated as failed block on dermatomal examination after block application

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-85 years who underwent surgery for femoral neck fracture and underwent PENG block
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Numeric Rating Scale (NRS) | Postoperative 0th, 6th,12th and 24th hours
  Changes in Numeric Rating Scale (NRS) at rest and in activity will be recorded at intervals. At 0-6-12-24 hours, pain will be evaluated with the NRS score in two different situations.
  Patients will be informed about the Numeric Rating Scale used in the assessment of pain and pain intensity will be determined at rest and 24 hours postoperatively during 15 degrees passive leg raising. Patients will be asked to express their pain intensity numerically between 0 and 10, with 0 for no pain and 10 for the most severe pain.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | Postoperative 6th, 12th and 24th hours
  The severity of nausea and vomiting was determined by a four-point Verbal Descriptive Scale.
The degree of motor block | Postoperative 6th, 12th and 24th hours
  The degree of motor block will be evaluated with the Bromage scale.
The degree of sensory block | Postoperative 6th, 12th and 24th hours
  The degree of sensory block will be evaluated with the Pinprick test.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kelsaka, Prof.Dr, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Maxwell MJ, Moran CG, Moppett IK. Development and validation of a preoperative scoring system to predict 30 day mortality in patients undergoing hip fracture surgery. Br J Anaesth. 2008 Oct;101(4):511-7. doi: 10.1093/bja/aen236. Epub 2008 Aug 21. PMID 18723517
- [Background] Abou-Setta AM, Beaupre LA, Rashiq S, Dryden DM, Hamm MP, Sadowski CA, Menon MR, Majumdar SR, Wilson DM, Karkhaneh M, Mousavi SS, Wong K, Tjosvold L, Jones CA. Comparative effectiveness of pain management interventions for hip fracture: a systematic review. Ann Intern Med. 2011 Aug 16;155(4):234-45. doi: 10.7326/0003-4819-155-4-201108160-00346. PMID 21844549
- [Background] Parker MJ, Handoll HH, Griffiths R. Anaesthesia for hip fracture surgery in adults. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD000521. doi: 10.1002/14651858.CD000521.pub2. PMID 15494999
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271